CLINICAL TRIAL: NCT00203372
Title: A Multicenter, Placebo-Controlled, Double-Blind Randomized Phase II Trial of Neoadjuvant Treatment With Single-Agent Bevacizumab or Placebo, Followed by Six Cycles of Docetaxel, Doxorubicin, and Cyclophosphamide (TAC), With or Without Bevacizumab in Patients With Stage II or Stage III Breast Cancer
Brief Title: Neoadjuvant TAC Plus or Minus Bevacizumab(AVF3299)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Translational Oncology Research International (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TORI B-02; 10-001419 (Other: JCCC IRB); NCT00128674 (obsolete NCT alias)
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2011-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Docetaxel; Doxorubicin; Cyclophosphamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Bevacizumab 7.5 and TAC (Experimental): one dose of Bevacizumab (7.5mg/kg) will be administered intravenously every 3 weeks followed by TAC.
  Interventions: Drug: Bevacizumab 7.5 and TAC
- Placebo 7.5 and TAC (Placebo Comparator): Placebo7.5 will be administered intravenously every 3 weeks followed by TAC.
  Interventions: Drug: Placebo 7.5 and Docetaxel, Doxorubicin, and Cyclophosphamide (TAC)
- Bevacizumab 15 and TAC (Experimental): one dose of Bevacizumab (15mg/kg) will be administered intravenously every 3 weeks followed by TAC.
  Interventions: Drug: Bevacizumab 15 and TAC
- Placebo 15 and TAC (Placebo Comparator): Placebo 15mg/kg will be administered intravenously every 3 weeks followed by TAC.
  Interventions: Drug: Placebo 15 and TAC

INTERVENTIONS:
Drug: Bevacizumab 7.5 and TAC — Bevacizumab given intravenously at a dose of 7.5mg/kg every 3 weeks, followed by docetaxel, doxorubicin and cyclophosphamide (TAC).
  Arms: Bevacizumab 7.5 and TAC
Drug: Placebo 7.5 and Docetaxel, Doxorubicin, and Cyclophosphamide (TAC) — placebo 7.5 will be adminitered intravenously every 3 weeks followed by TAC
  Arms: Placebo 7.5 and TAC
Drug: Bevacizumab 15 and TAC — one dose of Bevacizumab (15 mg/kg) will be administered intravenously every 3 weeks followed by TAC.
  Arms: Bevacizumab 15 and TAC
Drug: Placebo 15 and TAC — one dose of placebo 15 will be administered intravenously every 3 weeks followed by TAC.
  Arms: Placebo 15 and TAC

SUMMARY:
The purpose of this study is to evaluate the safety of the TAC-bevacizumab combination and investigate whether changes in gene expression, or the expression of specific biomarkers, are either predictive of response to bevacizumab or indicative of response.

DETAILED DESCRIPTION:
The study combines bevacizumab with a very efficacious combination chemotherapy regimen for the treatment of stage II or stage III primary breast cancer. Safety of the TAC-bevacizumab combination will be evaluated. In addition, the study design incorporates an initial cycle of bevacizumab or placebo alone. Assessing the isolated effects of bevacizumab in a setting where pre- and post-treatment tissue specimens can be obtained will provide essential information about the mechanisms by which VEGF inhibition affects tumor growth, and represents an ideal opportunity to evaluate the molecular effects of bevacizumab on breast tumor tissue.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proven adenocarcinoma of the breast
* Stage II (T > 3 cm) or Stage III disease (except inflammatory breast cancer), according to the AJCC Staging Manual, 6th Edition, 2002
* HER2-negative disease (as defined by fluorescence in situ hybridization [FISH])
* ECOG performance status 0-1
* No prior chemotherapy, radiotherapy, or endocrine therapy for invasive or noninvasive breast cancer
* Normal cardiac function (ejection fraction > lower limit of normal) as determined by MUGA or echocardiogram
* Adequate organ function

Exclusion Criteria:

* Prior chemotherapy or radiotherapy for Stage II or Stage III breast cancer
* Inflammatory Breast Cancer, clinically defined as the presence of erythema or induration involving one-third or more of the breast
* Prior treatment with an anti-angiogenic agent
* Prior ipsilateral radiation therapy for invasive or non-invasive breast cancer
* Bilateral invasive breast cancer
* Concurrent therapy with any other non-protocol anti-cancer therapy
* Current therapy with hormone replacement therapy, or any hormonal agent such as raloxifene, tamoxifen, or other selective estrogen receptor modulators (agents must be stopped prior to randomization)
* Presence of neuropathy > grade 2 (NCI-CTC version 3.0) at baseline
* Presence of any non-healing wound, bone fracture, or ulcer, or the presence of clinically significant (> grade 2) peripheral vascular disease
* History of any other malignancy within the past 5 years, with the exception of non-melanoma skin cancer or carcinoma-in-situ of the cervix
* Clinically significant cardiovascular disease (e.g., hypertension [BP > 150/100], myocardial infarction or stroke within 6 months, unstable angina), New York Heart Association (NYHA) Grade II or greater congestive heart failure, or serious cardiac arrhythmia requiring medication
* Active peptic ulcer disease, inflammatory bowel disease, or other gastrointestinal condition increasing the risk of perforation; history of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to beginning therapy
* Active, uncontrolled infection requiring parenteral antimicrobials
* The presence of any other medical or psychiatric disorder that, in the opinion of the treating physician, would contraindicate the use of the drugs in this protocol or place the subject at undue risk for treatment complications
* Pregnancy or lactation
* A history of a severe hypersensitivity reaction to bevacizumab, or docetaxel or other drugs formulated with polysorbate 80
* Evidence of bleeding diathesis or coagulopathy
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to beginning therapy, or anticipation of the need for a major surgical procedure during the course of the study; minor surgical procedure, fine needle aspiration, or core biopsy within 7 days prior to beginning therapy
* Urine protein:creatinine ratio of > 1.0 at screening

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2005-05; Primary Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
•To evaluate the safety and toxicity of the TAC regimen with the addition of bevacizumab given as preoperative therapy to patients with Stage II or Stage III breast cancer | 4 years
  Patients will be evaluated for adverse events (all grades) at each study visit for the duration of their participation in the study. All AEs should be graded using the NCI--CTCAE, Version 3.0. Patients discontinued from the treatment phase of the study for any reason will be evaluated within 30 days after the decision to discontinue treatment.
•To estimate change from baseline expression of HIF1α as a measure of tumor angiogenesis, after a single dose of bevacizumab as compared to placebo | 4 years

SECONDARY OUTCOMES:
•To estimate the rate of CHF in patients receiving TAC with or without bevacizumab | 4 years
•To estimate the rates of left ventricular ejection fraction (LVEF) changes as measured by either a decrease of > 15% from baseline, or > 10% to a value below the lower limit of normal (for the institution), in patients receiving TAC or TAC + bevacizumab | 4 years
•To investigate the clinical efficacy of TAC and TAC plus bevacizumab by estimating the clinical objective response rate (CR + PR), pathologic complete response rate (pCR), and rate of breast-conserving surgery (BCS) | 4 years
•To estimate the rate of post-surgical wound healing complications in patients who receive surgery after TAC or TAC plus bevacizumab | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Fairooz Kabbinavar, MD, Study Chair — Chief Medical Officer
Locations (9):
- United States (5):
  - UCLA Medical Center, Los Angeles, California
  - Wilshire Oncology Medical Group, Inc., Pomona, California
  - Cancer Institute of Florida, P.A., Orlando, Florida
  - Northwest Georgia Oncology Centers, P.C., Marietta, Georgia
  - South Texas Oncology and Hematology, P.A., San Antonio, Texas
- Canada (2):
  - Cross Cancer Institute, Edmonton, Alberta
  - McGill University, Montreal, Quebec
- Ireland (2):
  - St. Vincent's University Hospital, Dublin
  - St. James's Hospital, Dublin